CLINICAL TRIAL: NCT07225660
Title: A Randomized Blinded Controlled Trial Assessing Hormonal Optimization: Late vs. Immediate Start After Discontinuation of Oral Contraceptives in Assisted Reproductive technologY (HOLIDAY)
Acronym: HOLIDAY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shady Grove Fertility Reproductive Science Center (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Kate Devine, Medical Director and Chief Research Officer, USFertility, Shady Grove Fertility Reproductive Science Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00090115
Record Dates: First submitted 2025-11-04; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Fertility Preservation
Keywords: planned oocyte cryopreservation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holiday (Other): Patients will undergo a 2 month drug holiday (pause) with combined hormonal contraceptives prior to planned oocyte cryopreservation
  Interventions: Other: OCP pause
- Immediate Start (No Intervention): Patients will immediately begin planned oocyte cryopreservation after discontinuation of prolonged combined hormonal contraceptive

INTERVENTIONS:
Other: OCP pause — Subjects in the study arm will be asked to discontinue combined hormonal contraceptives (CHC) for 2 months prior to planned oocyte cryopreservation
  Arms: Holiday

SUMMARY:
HOLIDAY is a two-arm, parallel-group, multi-center, randomized trial in which subjects undergoing planned oocyte cryopreservation will be randomized to receive either a 2-month pause of Combined Hormonal Contraceptives (CHC) or immediate start (without a pause).

DETAILED DESCRIPTION:
Reproductive aging in women is a continuous process that begins prior to birth and extends until menopause. The primary mechanism behind this process is the depletion of the ovarian pool of non-growing follicles (NGFs). Previous models, such as the biphasic-exponential model [1], have postulated that female fertility prominently declines with age, significantly after age 32, and with a more accelerated rate after age 35 [2,3]. Newer models of ovarian follicular depletion predict no sudden change in decay rate but rather a constantly, increasing rate [4].

With the advent of vitrification [5], oocyte cryopreservation has become a powerful tool to help preserve female fertility potential against anticipated gamete exhaustion. At the same time, as more women choose to delay childbearing for various reasons, planned oocyte preservation is increasing in popularity [6-8]. Continued optimization of protocols has led to improved outcomes with good oocyte yields [9]. For women undergoing oocyte cryopreservation who are not actively attempting to conceive, endometrial development does not need to be synchronized with the oocytes. Thus, ovarian stimulation can be initiated irrespective of the phase of the menstrual cycle without adversely impacting oocyte yield or quality, thereby facilitating scheduling and reducing delays [10].

Many patients are utilizing combined hormonal contraception (CHC) at the time of their initial oocyte cryopreservation consultation [11]. In the United States, about 14% of women aged 15-49 were using oral contraceptive pills (OCPs) in 2017-2019 [12]. While a short course of CHC exposure is unlikely to be detrimental to oocyte yield [13-15], longer-term CHC use may lead to significant suppression of the hypothalamic-pituitary-ovarian axis, gonadotropins, and in turn, follicular development. After only 3 months of CHC use, studies have demonstrated that the pituitary response to gonadotropin-releasing hormone is blunted [16-18]. If hypothalamic-pituitary suppression from CHC prevents progression of follicle development to the antral stage, prolonged use may also lower the number of follicles susceptible to exogenous gonadotropin stimulation for oocyte collection and therefore total oocyte yield. Patients may require additional cycles and incur additional expense to achieve the desired number of cryopreserved oocytes.

It has been well demonstrated that markers of ORT [19], specifically, antral follicle count (AFC) and Anti-Müllerian hormone (AMH) are good predictors of oocyte yield [20-22]. Existing evidence suggests that CHC use can suppress and diminish these measures of ovarian reserve by 20-30% [23-24] via suppression of follicle-stimulating hormone (FSH). One study found that that long-term CHC user could increase AMH by 53% and AFC by 41%, with values returning to normal within 2 months and a plateau effect thereafter [25]. Similarly, another study found after stopping long-term CHC use for 2 months, there was an average increase in AFC of 4 [26].

Overall, existing literature regarding the association between hormonal contraceptive use and AMH concentration has historically been inconsistent [27-31] but more recent data with large sample sizes [33], including a systematic review, concluded that AMH levels in women using CHC more than 6 months appears to markedly decline with recovery after discontinuation [34]. Reproductive-age women with lower AMH percentiles at baseline may experience a greater suppressive effect from prolonged CHC use, while it is speculated that those with higher AMH percentiles at baseline may experience a lesser suppressive effect [35].

There are abundant observational data suggesting long-term CHC use is associated with reversable suppression of ovarian reserve markers, with biologic plausibility that this in turn may mask the "true biological potential" of the ovaries and possibly result in suboptimal oocyte yield. However, to date there are no published adequately powered prospective randomized data evaluating whether a contraceptive pause would lead to improved outcomes. Such practices may already be taking place in ART centers. The simple act of waiting for the potential of more oocytes takes on an obvious, low-risk appeal. Therefore, we propose this assessor-blind, randomized clinical trial comparing a 2-month contraceptive pause to immediate oocyte cryopreservation, with oocyte yield as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Ovary-bearing individuals 18 to 40 years of age.
2. BMI < 40 kg/m2
3. Non-smoker for at least 3 months prior to study enrollment.

Exclusion Criteria:

1. BMI greater than or equal to 40 kg/m2
2. Current Smoker
3. Any contraindications to ovarian stimulation or outpatient egg retrieval under anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 394 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Oocyte maturation rate | During oocyte retrieval
  Median number of percentage of vitrified MII oocytes yielded per cycle
Number of oocytes retrieved | During oocyte retrieval
  The median number of cumulus-oocyte complexes (COC) retrieved during oocyte retrieval

SECONDARY OUTCOMES:
AMH levels | AMH level differences from baseline to post-drug holiday (2 months)
  Differences in AMH levels from baseline to cycle start

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Yale Fertility Center, Orange, Connecticut
  - Shady Grove Fertility Rockville, Rockville, Maryland
  - Reproductive Medicine Associates of New York, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen BL, Katz M. Further studies on pituitary and ovarian function in women receiving hormonal contraception. Contraception. 1981 Aug;24(2):159-72. doi: 10.1016/0010-7824(81)90089-5. PMID 6794980
- [Background] Wan LS, Ganguly M, Weiss G. Pituitary response to LHRH stimulation in women on oral contraceptives: a followup dose response study. Contraception. 1981 Sep;24(3):229-34. doi: 10.1016/0010-7824(81)90035-4. PMID 6796328
- [Background] Yu Ng EH, Chi Wai Chan C, Tang OS, Shu Biu Yeung W, Chung Ho P. Effect of pituitary downregulation on antral follicle count, ovarian volume and stromal blood flow measured by three-dimensional ultrasound with power Doppler prior to ovarian stimulation. Hum Reprod. 2004 Dec;19(12):2811-5. doi: 10.1093/humrep/deh500. Epub 2004 Sep 9. PMID 15358718
- [Background] Tran ND, Aghajanova L, Kao CN, Cedars MI, Rosen MP. Impact of pituitary suppression on antral follicle count and oocyte recovery after ovarian stimulation. Fertil Steril. 2016 Mar;105(3):690-696. doi: 10.1016/j.fertnstert.2015.11.033. Epub 2015 Dec 13. PMID 26696299
- [Background] Cohen BL, Katz M. Pituitary and ovarian function in women receiving hormonal contraception. Contraception. 1979 Nov;20(5):475-87. doi: 10.1016/0010-7824(79)90053-2. PMID 393456
- [Background] Daniels K, Abma JC. Current Contraceptive Status Among Women Aged 15-49: United States, 2017-2019. NCHS Data Brief. 2020 Oct;(388):1-8. PMID 33151146
- [Background] Schattman GL. Cryopreservation of Oocytes. Author replies. N Engl J Med. 2016 Jan 21;374(3):288. doi: 10.1056/NEJMc1515128. No abstract available. PMID 26789885
- [Background] Doyle JO, Richter KS, Lim J, Stillman RJ, Graham JR, Tucker MJ. Successful elective and medically indicated oocyte vitrification and warming for autologous in vitro fertilization, with predicted birth probabilities for fertility preservation according to number of cryopreserved oocytes and age at retrieval. Fertil Steril. 2016 Feb;105(2):459-66.e2. doi: 10.1016/j.fertnstert.2015.10.026. Epub 2015 Nov 18. PMID 26604065
- [Background] Cil AP, Bang H, Oktay K. Age-specific probability of live birth with oocyte cryopreservation: an individual patient data meta-analysis. Fertil Steril. 2013 Aug;100(2):492-9.e3. doi: 10.1016/j.fertnstert.2013.04.023. Epub 2013 May 24. PMID 23706339
- [Background] Mesen TB, Mersereau JE, Kane JB, Steiner AZ. Optimal timing for elective egg freezing. Fertil Steril. 2015 Jun;103(6):1551-6.e1-4. doi: 10.1016/j.fertnstert.2015.03.002. Epub 2015 Apr 14. PMID 25881876
- [Background] Rudick B, Opper N, Paulson R, Bendikson K, Chung K. The status of oocyte cryopreservation in the United States. Fertil Steril. 2010 Dec;94(7):2642-6. doi: 10.1016/j.fertnstert.2010.04.079. Epub 2010 Jun 18. PMID 20723535
- [Background] Noyes N, Porcu E, Borini A. Over 900 oocyte cryopreservation babies born with no apparent increase in congenital anomalies. Reprod Biomed Online. 2009 Jun;18(6):769-76. doi: 10.1016/s1472-6483(10)60025-9. PMID 19490780
- [Background] Hansen KR, Knowlton NS, Thyer AC, Charleston JS, Soules MR, Klein NA. A new model of reproductive aging: the decline in ovarian non-growing follicle number from birth to menopause. Hum Reprod. 2008 Mar;23(3):699-708. doi: 10.1093/humrep/dem408. Epub 2008 Jan 11. PMID 18192670
- [Background] Sozou PD, Hartshorne GM. Time to pregnancy: a computational method for using the duration of non-conception for predicting conception. PLoS One. 2012;7(10):e46544. doi: 10.1371/journal.pone.0046544. Epub 2012 Oct 4. PMID 23056338
- [Background] Dunson DB, Baird DD, Colombo B. Increased infertility with age in men and women. Obstet Gynecol. 2004 Jan;103(1):51-6. doi: 10.1097/01.AOG.0000100153.24061.45. PMID 14704244
- [Background] Faddy MJ, Gosden RG, Gougeon A, Richardson SJ, Nelson JF. Accelerated disappearance of ovarian follicles in mid-life: implications for forecasting menopause. Hum Reprod. 1992 Nov;7(10):1342-6. doi: 10.1093/oxfordjournals.humrep.a137570. PMID 1291557